CLINICAL TRIAL: NCT06216197
Title: Dexmedetomidine Versus Fentanyl as an Adjuvant to Bupivacaine in Saddle Block for Various Anal Surgeries: A Correlative Randomized Trial
Brief Title: Dexmedetomidine Versus Fentanyl as an Adjuvant to Bupivacaine in Saddle Block
Acronym: saddle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zulekha Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 0395/2023
Record Dates: First submitted 2023-12-26; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Regional Anesthesia Morbidity

STUDY DESIGN:
Intervention Model Description: Fifty-eight adult patients were categorized into two groups. Group FENT, consisting of 29 patients, underwent a saddle block with hyperbaric bupivacaine (2.5 ml) combined with fentanyl (0.5 ml; 25 μg). The DEX Group, consisting of 29 patients, received 2.5 ml of hyperbaric bupivacaine mixed with dexmedetomidine (10 μg; 0.5 ml).
Who Masked: Investigator
Masking Description: The subjects were randomly categorized into two groups utilizing random numbers generated by computer software. A sealed envelope (containing the allocation numbers of groups) was opened at the time of patient enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The FENT Group (Other): Group FENT, consisting of 29 patients, underwent a saddle block with hyperbaric bupivacaine (2.5 ml) combined with fentanyl (0.5 ml; 25 μg).
  Interventions: Drug: FENT group
- The DEX Group (Other): The DEX Group, consisting of 29 patients, received 2.5 ml of hyperbaric bupivacaine mixed with dexmedetomidine (10 μg; 0.5 ml).
  Interventions: Drug: DEX group

INTERVENTIONS:
Drug: FENT group — Group FENT, consisting of 29 patients, underwent a saddle block with hyperbaric bupivacaine (2.5 ml) combined with fentanyl (0.5 ml; 25 μg).
  Other Names: fentanyl group
  Arms: The FENT Group
Drug: DEX group — The DEX Group, consisting of 29 patients, received 2.5 ml of hyperbaric bupivacaine mixed with dexmedetomidine (10 μg; 0.5 ml).
  Other Names: dexmedetomidine group
  Arms: The DEX Group

SUMMARY:
Dexmedetomidine is recommended over fentanyl as adjunctive medication to bupivacaine for saddle block spinal anesthesia in anal surgeries and procedures.

DETAILED DESCRIPTION:
Objectives: A saddle spinal block is a viable choice for anal surgeries. This technique effectively maintains balanced hemodynamics, and fast recovery, and prevents irrelevant motor blocks in both limbs.

Methods: Fifty-eight adult patients were categorized into two groups. Group FENT, consisting of 29 patients, underwent a saddle block with hyperbaric bupivacaine (2.5 ml) combined with fentanyl (0.5 ml; 25 μg). The DEX Group, consisting of 29 patients, received 2.5 ml of hyperbaric bupivacaine mixed with dexmedetomidine (10 μg; 0.5 ml). Continuous monitoring of HR and SpO2 was conducted. Evaluation of sensory blockage and the motor block was done utilizing the Bromage scale. Following surgery, assessments were conducted. Pain in the ward and PACU was determined utilizing the visual analog scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* aged between 20 and 60
* classified as II & ASA-I
* scheduled for elective anal surgeries

Exclusion Criteria:

* subjects who refused to participate
* uncontrolled hypertension
* BMI > 30 kg/m2
* heart failure (class IV or III) based on the New York Heart Association (NYHA)
* uncorrected coagulopathy
* any study's drug allergy
* drug abuse
* neuropathy
* any spinal anesthesia contraindication (such as infection or a pelvic fracture)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2021-04-03 (Actual); Primary Completion 2022-12-04 (Actual); Study Completion 2022-12-04 (Actual)

PRIMARY OUTCOMES:
the duration until the first call for analgesia | 20 months
  the duration until the first call for analgesia

SECONDARY OUTCOMES:
the duration from spinal injection until reaching the maximal sensory level | 20 months
  the duration from spinal injection until reaching the maximal sensory level
the duration needed for sensory regression to occur over two spinal segments from the maximal sensory level | 20 months
  the duration needed for sensory regression to occur over two spinal segments from the maximal sensory level
the time required for sensory regression until reaching the S1 level (from the maximal sensory level) | 20 months
  the time required for sensory regression until reaching the S1 level (from the maximal sensory level)
the duration from injection to achieving Bromage 0, the total tramadol consumption (until the first 24 hours) | 20 months
  the duration from injection to achieving Bromage 0, the total tramadol consumption (until the first 24 hours)
side effects occurrences | 20 months
  side effects occurrences

CONTACTS AND LOCATIONS:
Overall Officials: sameh ha seyam, MD, Study Chair — assistant professor of anesthesiology, intensive care and pain management
Locations (1):
- Al-Azhar faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
available